CLINICAL TRIAL: NCT06419361
Title: [68Ga]Ga-Sa-DABI-4 PET Imaging of Stimulator of Interferon Gene Expression in Cancer Patients
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: First Affiliated Hospital of Chongqing Medical University (Other)
Responsible Party: Principal Investigator, Xiaoyang Zhang, Principal Investigator, First Affiliated Hospital of Chongqing Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CYYY-KY-2024-049-01
Record Dates: First submitted 2024-05-14; First posted 2024-05-17 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-05

CONDITIONS: Stimulator of Interferon Gene; Cancer; Positron Emission Tomography
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- [68Ga]Ga-Sa-DABI-4 (Experimental): Patients will receive a single administration of [68Ga]Ga-Sa-DABI-4.
  Interventions: Drug: [68Ga]Ga-Sa-DABI-4

INTERVENTIONS:
Drug: [68Ga]Ga-Sa-DABI-4 — Each subject receives a single intravenous injection of [68Ga]Ga-Sa-DABI-4.

SUMMARY:
Stimulator of interferon gene (STING) protein plays a vital role in the immune surveillance of tumor microenvironment. Monitoring STING expression in tumors benefits the relevant STING therapy. This study will investigate the safety, biodistribution and potential usefulness of a novel 68Ga-labeled agonist ([68Ga]Ga-Sa-DABI-4) for noninvasive positron emission tomography (PET) imaging of STING expression in the tumor microenvironment.

ELIGIBILITY:
Inclusion Criteria:

1. At least 18 years of age.
2. Signed informed consent.
3. Patients with suspected or newly diagnosed or previously malignant disease.

Exclusion Criteria:

1. Patients with non-malignant disease.
2. Patients with pregnancy.
3. The inability or unwillingness of the research participant, parent or legal representative to provide written informed consent.
4. Known or expected hypersensitivity to [68Ga]Ga-Sa-DABI-4 or any of its components.
5. Any serious medical condition or extenuating circumstance which the investigator feels may interfere with the procedures or evaluations of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-05-30 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Diagnostic efficacy | 15 days
  The sensitivity, specificity, and accuracy of [68Ga]Ga-Sa-DABI-4 PET

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: No